CLINICAL TRIAL: NCT02696967
Title: A Randomized, Subject and Investigator-blind, Placebo-controlled Study of CLR325 in Chronic Stable Heart Failure Patients
Brief Title: A Study of CLR325 in Chronic Stable Heart Failure Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCLR325X2202; 2016-001387-12 (EudraCT Number)
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-09

CONDITIONS: Chronic Stable Heart Failure
Keywords: Apelin; CLR325; Chronic heart failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLR325 (Experimental): Patients were assigned to one of the 2 treatment arms in fixed randomization ratio. Patients randomized to this arm received single dose of CLR325 (i.v.) in double blind manner.
  Interventions: Drug: CLR325
- Placebo (Placebo Comparator): Patients were assigned to one of the 2 treatment arms in fixed randomization ratio. Patients randomized to this arm received single dose of placebo (i.v.) in double blind manner.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CLR325 — CLR325 Concentrate for solution for infusion
  Arms: CLR325
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the safety and tolerability of CLR325 intravenous (i.v.) infusion in patients with stable heart failure to determine if further clinical development of the drug in this indication was warranted.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients >18 years of age
* Body weight between 50 kg and 140 kg
* Cardiac ejection fraction of ≤ 45% assessed within the last 6 months
* For PA catheter cohorts, patients who are planned to have a clinically indicated pulmonary artery catheter in place prior to randomization
* In the opinion of the investigator, heart failure patients who do not require a change in their dose of acetylcholinesterase (ACE), angiotensin receptor blocker (ARB), β-blocker, mineralocorticoid receptor antagonist, or diuretic for 24 h after randomization.
* At Baseline, vital signs (systolic and diastolic blood pressure and pulse rate) assessment in the supine position after the subject has rested for at least five minutes.

Key Exclusion Criteria:

* Impaired renal function as indicated by clinically significant abnormal creatinine values (Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 calculated using the Modification of Diet in Renal Disease Study (MDRD) equation)
* History of chronic hepatitis of any non-cardiac etiology
* History of any active or clinically significant cardiac tachyarrhythmia (such as recurrent atrial fibrillation with rapid ventricular response within the last year) and patients with chronic atrial fibrillation with a pulse rate ≤ 100 bpm
* Patients who received an i.v. infusion of a cardiac inotrope (e.g., dobutamine or milrinone) in the last 24 h prior to randomization
* Patients with any significant change in their dose of their ACE, ARB, mineralocorticoid receptor antagonist, diuretic, or β-blocker within the last 12 h
* Patients with known significant valvular heart diseases indicated by the following:

  * severe aortic stenosis (aortic valve area < 1.0 cm2 or peak gradient > 50 mm Hg as determined by echocardiography)
  * severe mitral stenosis
* History of acute coronary syndrome within the last 60 days as determined by both clinical and enzymatic criteria
* For echocardiography-based cohorts only, patients admitted to an inpatient setting for acute decompensated heart failure within the last 30 days
* For PA catheter cohorts, patients with a pulmonary capillary wedge pressure of <10 mm Hg at Baseline. For echocardiographic cohorts, patients with a lateral E/E' ratio of < 7 on their baseline echocardiogram. For patients in whom a lateral E/E' ratio cannot be determined (e.g., patients in atrial fibrillation), a central venous pressure of < 5 mm Hg on baseline echocardiogram as determined by inferior vena cava criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (6):
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Tacoma, Washington
- Novartis Investigative Site, Aalst, Belgium
- Germany (2):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Greifswald
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 11 centers in 5 countries: Belgium (1), Germany (2), Netherlands (1), Singapore (1) and USA (6).
Pre-assignment Details: Patients were assigned to one of the 2 treatment arms in fixed randomization ratio (CLR325: Placebo):
  * Cohort 1: Single dose of CLR325 2.5 mcg/kg/min (i.v.) or placebo (i.v.)
  * Cohort 2: Single dose of CLR325 0.25 mcg/kg/min (i.v.) or placebo (i.v.)
  * Cohort 3: Single dose of CLR325 8 mcg/kg/min (i.v.) or placebo (i.v.)
Groups:
- CLR325 0.25 mcg/kg/Min: Patients randomized to this arm received single dose of CLR325 0.25 mcg/kg/min (i.v.) in double blind manner.
- CLR325 2.5 mcg/kg/Min: Patients randomized to this arm received single dose of CLR325 2.5 mcg/kg/min (i.v.) in double blind manner.
- CLR325 8 mcg/kg/Min: Patients randomized to this arm received single dose of CLR325 8 mcg/kg/min (i.v.) in double blind manner.
- Placebo: Patients randomized to this arm received single dose of Placebo (i.v.) in double blind manner.
Period: Overall Study
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min | Placebo
Started (All randomized patients were included in the Full Analysis Set (FAS) and Safety Analysis Set (SAF).) | 4 | 6 | 6 | 10
Pharmacokinetic (PK) Analysis Set (At least one dose of study drug and one evaluable PK concentration measurement) | 4 | 6 | 4 | 0
Completed | 4 | 6 | 6 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min | Placebo | Total
Number analyzed (Participants) | 4 | 6 | 6 | 10 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (3.1) | 55.2 (13.0) | 63.5 (11.8) | 54.2 (9.2) | 56.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 0 | 3
  Male | 3 | 6 | 4 | 10 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 4 | 3 | 4 | 8 | 19
  Black | 0 | 2 | 2 | 1 | 5
  Asian | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death
Description: Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) in each treatment arm to demonstrate that CLR325 is safe for the treatment of chronic stable heart-failure patients through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: Day 1 to 28
Population: The Safety population, which consisted of all patients who had been exposed to at least one infusion of study drug or placebo, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min | Placebo
Number analyzed (Participants) | 4 | 6 | 6 | 10
Participants
  On-treatment Adverse Event (AEs) | 1 | 2 | 4 | 7
  On-treatment Serious Adverse Event (SAEs) | 0 | 2 | 2 | 0
  On-treatment Deaths | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Area Under the Plasma Concentration-time Curve From Time Zero to 18 Hours (AUC0-18hr)
Description: AUC0-18hr is the area under the plasma concentration-time curve from time zero to 18 hours after the start of CLR325 infusion. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0, 0.5, 3, 5, 8, 10, 12, and 18 hours post start of CLR325 infusion on Day 1
Population: Participants from the Pharmacokinetic (PK) analysis set, defined as all randomized participants who received at least one dose of study drug and one evaluable PK concentration measurement, with data available for analysis were considered.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
ng*hr/mL
  CLR 325 | 1220 (10.4) | 18500 (31.6) | 79700 (32.5)
  CQJ295 | NA (NA) — N/A: Not Estimable (CQJ295 concentration below lower limit of quantification (LLOQ)) | 623 (102.3) | 5560 (46.7)

3. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Area Under the Plasma Concentration-time Curve From From Time Zero to 28 Hours (AUC0-28hrs)
Description: AUC0-28hr is the area under the plasma concentration-time curve from time zero to 28 hours after the start of CLR325 infusion. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0, 0.5, 3, 5, 8, 10, 12, 18, 20, 24, and 28 hours post start of CLR325 infusion on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
ng*hr/mL
  CLR325 | 1460 (12.8) | 21500 (32.9) | 100000 (28.2)
  CQJ295 | NA (NA) — N/A: Not Estimable (CQJ295 concentration below lower limit of quantification (LLOQ)) | 838 (106.2) | 8390 (43.5)

4. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: AUCinf is the area under the plasma concentration-time curve from time zero to infinity. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0, 0.5, 3, 5, 8, 10, 12, 18, 20, 24, and 28 hours post start of CLR325 infusion on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 2 | 6 | 4
ng*hr/mL
  CLR325 | 1510 (4.7) | 21900 (34.0) | 103000 (26.1)
  CQJ295: number analyzed (Participants) | 0 | 4 | 4
  CQJ295 |  | 843 (49.9) | 9660 (38.5)

5. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Description: AUClast is the area under the plasma concentration-time curve from time zero to the last measurable concentration sampling time. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0, 0.5, 3, 5, 8, 10, 12, 18, 20, 24, and 28 hours post start of CLR325 infusion on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
ng*hr/mL
  CLR325 | 1450 (13.0) | 21500 (32.9) | 100000 (28.2)
  CQJ295: number analyzed (Participants) | 1 | 6 | 4
  CQJ295 | 3.10 (NA) — NA: Not estimable due to insufficient number of participants with events | 836 (107.1) | 8380 (43.6)

6. Secondary Outcome: Pharmacokinetic of CLR325: Clearance From Plasma (CL) Following Drug Administration
Description: CL is the systemic (or total body) clearance from plasma following CLR325 infusion. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0, 0.5, 3, 5, 8, 10, 12, 18, 20, 24, and 28 hours post start of CLR325 infusion on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
mL/hr | 15200 (6.1) | 13200 (54.9) | 7460 (15.4)

7. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax,ss)
Description: Cmax,ss is the observed maximum plasma concentration following drug administration at steady state. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0, 0.5, 3, 5, 8, 10, 12, 18, 20, 24, and 28 hours post start of CLR325 infusion on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
ng/mL
  CLR325 | 103 (11.2) | 1370 (36.0) | 6080 (38.4)
  CQJ295 | NA (NA) — N/A: Not Estimable (CQJ295 concentration below lower limit of quantification (LLOQ)) | 54.2 (91.0) | 468 (54.0)

8. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Terminal Elimination Half-life (T1/2)
Description: T^1/2 is the elimination half-life associated with the terminal slope of a semi logarithmic concentration-time curve. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 18, 20, 24, and 28 hours post start of CLR325 infusion on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 2 | 6 | 4
hr
  CLR325 | 1.86 (0.197) | 2.99 (0.520) | 2.96 (0.992)
  CQJ295: number analyzed (Participants) | 0 | 4 | 4
  CQJ295 |  | 3.12 (0.275) | 5.73 (3.38)

9. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Time to Reach the Maximum Concentration After Drug Administration (TMax)
Description: Tmax is the time to reach maximum plasma concentration after single dose administration. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0, 0.5, 3, 5, 8, 10, 12, 18, 20, 24, and 28 hours post start of CLR325 infusion on Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
hr
  CLR325 | 14.0 [4.93 to 18.0] | 12.0 [8.05 to 12.1] | 14.9 [8.08 to 17.9]
  CQJ295 | 0 [0 to 5.03] | 15.1 [7.92 to 18.1] | 17.9 [8.33 to 18.1]

10. Secondary Outcome: Pharmacokinetic of CLR325: Volume of Distribution at Steady State Following Intravenous Administration (Vss)
Description: Vss is the volume of distribution at steady state following intravenous administration. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0, 0.5, 3, 5, 8, 10, 12, 18, 20, 24, and 28 hours post start of CLR325 infusion on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
mL | 51600 (19.6) | 32500 (47.6) | 28000 (33.3)

11. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Amount of Drug (or Defined Metabolite) Excreted Into the Urine From Time (Ae 0-28 Hours)
Description: Ae 0-28 hours is the amount of drug (or defined metabolite) excreted into the urine from time zero to 28 hours after the start of CLR325 infusion. The urine PK parameters were measured using an non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0-28 hours on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
ng
  CLR325 | NA (NA) — N/A: Not Estimable (CLR325 concentration below lower limit of quantification (LLOQ)) | 19500000 (125.2) | 41300000 (253.3)
  CQJ295: number analyzed (Participants) | 3 | 4 | 1
  CQJ295 | NA (NA) — N/A: Not Estimable (CQJ295 concentration below lower limit of quantification (LLOQ)) | 7620000 (27.2) | 4040000 (NA) — NA: Not estimable due to insufficient number of participants with events

12. Secondary Outcome: Pharmacokinetic of CLR325 and CQJ295: Renal Clearance From Plasma (CLr) Following Drug Administration
Description: CLr is the renal clearance from urine following CLR325 infusion. The urine PK parameters were measured using an non-compartmental methods. Only descriptive analysis performed.
Time Frame: 0-28 hours on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min
Number analyzed (Participants) | 4 | 6 | 4
mL/hr
  CLR325: number analyzed (Participants) | 3 | 6 | 4
  CLR325 | NA (NA) — N/A: Not Estimable (CLR325 concentration below lower limit of quantification (LLOQ)) | 904 (199.4) | 411 (395.1)
  CQJ295: number analyzed (Participants) | 1 | 4 | 1
  CQJ295 | NA (NA) — N/A: Not Estimable (CQJ295 concentration below lower limit of quantification (LLOQ)) | 5620 (71.7) | 258 (NA) — NA: Not estimable due to insufficient number of participants with events

13. Secondary Outcome: Number of Patients With Increase in Anti-CLR325 and Anti-apelin Antibodies in Serum
Description: Anti-CLR325 anti-apelin antibodies in serum were analyzed predose, Day 10 and Day 28 to determine the immunogenicity of an 18-hour i.v. infusion of CLR325 in heart failure patients.
Time Frame: Baseline (BL), Day 10 (D10) and Day 28 (D28)
Population: The Safety population, which consisted of all patients who had been exposed to at least one infusion of study drug or placebo, was considered. Only subjest with or without anitbody detected were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min | Placebo
Number analyzed (Participants) | 4 | 6 | 6 | 10
Participants
  BL anti-Apelin antibody: number analyzed (Participants) | 1 | 1 | 1 | 0
  BL anti-Apelin antibody: Antibody detected = Yes | 0 | 0 | 0 | 0
  BL anti-Apelin antibody: Antibody detected = No | 1 | 1 | 1 | 0
  BL anti-CLR325 antibody: number analyzed (Participants) | 4 | 5 | 5 | 10
  BL anti-CLR325 antibody: Antibody detected = Yes | 0 | 0 | 0 | 0
  BL anti-CLR325 antibody: Antibody detected = No | 4 | 5 | 5 | 10
  D10 anti-Apelin antibody: number analyzed (Participants) | 0 | 0 | 1 | 1
  D10 anti-Apelin antibody: Antibody detected = Yes | 0 | 0 | 0 | 0
  D10 anti-Apelin antibody: Antibody detected = No | 0 | 0 | 1 | 1
  D10 anti-CLR325 antibody: number analyzed (Participants) | 3 | 4 | 6 | 7
  D10 anti-CLR325 antibody: Antibody detected = Yes | 0 | 0 | 0 | 0
  D10 anti-CLR325 antibody: Antibody detected = No | 3 | 4 | 6 | 7
  D28 anti-Apelin antibody: number analyzed (Participants) | 1 | 0 | 1 | 0
  D28 anti-Apelin antibody: Antibody detected = Yes | 0 | 0 | 0 | 0
  D28 anti-Apelin antibody: Antibody detected = No | 1 | 0 | 1 | 0
  D28 anti-CLR325 antibody: number analyzed (Participants) | 3 | 5 | 5 | 9
  D28 anti-CLR325 antibody: Antibody detected = Yes | 0 | 0 | 0 | 0
  D28 anti-CLR325 antibody: Antibody detected = No | 3 | 5 | 5 | 9

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose of study treatment until end of study treatment plus 30 days post-treatment, up to maximum duration of 1 month.
Description: All randomized patients received a single i.v. infusion of CLR325 or placebo for approximately 18 hours.
  Any sign or symptom that occurs during the study treatment and 30 days post-treatment follow up.
Arm/Group | CLR325 0.25 mcg/kg/Min | CLR325 2.5 mcg/kg/Min | CLR325 8 mcg/kg/Min | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/6 | 2/6 | 0/10
Other Adverse Events (participants affected / at risk) | 1/4 | 2/6 | 4/6 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLR325 0.25 mcg/kg/Min (N=4) | CLR325 2.5 mcg/kg/Min (N=6) | CLR325 8 mcg/kg/Min (N=6) | Placebo (N=10)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLR325 0.25 mcg/kg/Min (N=4) | CLR325 2.5 mcg/kg/Min (N=6) | CLR325 8 mcg/kg/Min (N=6) | Placebo (N=10)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Infusion site pruritus (General disorders) | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1
Pulmonary arterial wedge pressure decreased (Investigations) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT02696967/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT02696967/SAP_001.pdf